CLINICAL TRIAL: NCT03628976
Title: Noninvasive Vagus Nerve Stimulation (VNS) for Neuromotor Adaptations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia Institute of Technology (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: H18151; 1R03NS106088-01A1 (NIH)
Record Dates: First submitted 2018-08-08; First posted 2018-08-14 (Actual); Results first posted 2022-09-19 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-08

CONDITIONS: Healthy Young Adults
Keywords: tVNS, training, neuromotor adaptation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham-tVNS to ear lobe (Sham Comparator): Sham-tVNS will be applied to the ear lobe.
  Interventions: Other: tVNS; Other: Motor training
- tVNS to tragus (Active Comparator): tVNS will be applied to the tragus.
  Interventions: Other: tVNS; Other: Motor training

INTERVENTIONS:
Other: tVNS — Intervention
Other: Motor training — Same finger training for both arms

SUMMARY:
The study will examine how electrical stimulation of vagus nerve (i.e. nerve around the outer ear) from the skin surface during motor training influences a brain hormone (called norepinephrine), brain activity, and motor performance.

DETAILED DESCRIPTION:
Motor function is compromised with advanced age, and motor impairment is involved in various neuromotor injuries and disorders including stroke, spinal cord injury, amputation, and aging. Development of effective interventions for facilitating neuromotor adaptation is essential for accelerating or augmenting rehabilitation outcomes in the control of impaired limbs. The ultimate goal of the study is to find non-pharmacological and non-invasive neuromodulating interventions for enhancing the rehabilitation outcomes that may be applied to individuals with impaired motor function. In rats, implanted afferent vagus nerve stimulation paired with motor training enhanced neuromotor adaptation and motor recovery most likely through increased release of central neuromodulators that originate from the brainstem. The investigators propose to translate the findings in rats into humans by applying vagus nerve stimulation noninvasively. Transcutaneous VNS (tVNS) can noninvasively activate the brainstem including locus coeruleus, where norepinephrine (i.e. neuromodulator) is synthesized. However, it is unknown whether tVNS leads to increasing neuromodulators and facilitating neuromotor adaptations when combined with motor training in humans. With potential applicability of this novel intervention for facilitating neuromotor adaptation to various clinical human populations in future scope, it is essential to start with the basic understanding about the effect of tVNS on the neuromotor system and training-induced adaptation in neuromotor behavior in non-disabled humans. The overarching hypothesis is that an application of tVNS increases central norepinephrine and facilitates training-induced neuromotor adaptations in humans. The specific aim is to examine the effect of tVNS on central norepinephrine and training-induced neuromotor adaptations in humans. The effect of applying tVNS concurrently to visuomotor training will be investigated by comparing the changes in central norepinephrine and changes in the visuomotor skill and corticospinal excitability due to training with and without tVNS (sham) in non-disabled humans. The visuomotor skill will be assessed with the root-mean-square error of the produced force against the target force, which will be normalized to the maximal voluntary contraction force (MVC) . The investigators expect that subjects with concurrent tVNS during training show greater increases in the visuomotor skill and corticospinal excitability after training. The investigators also expect that tVNS increases central norepinephrine, and the amount of neuromotor adaptations due to training is associated with that of tVNS-induced increase in central norepinephrine. These expected findings will be the first evidence on the efficacy of concurrent tVNS with motor training for upregulating central norepinephrine and facilitating training-induced neuromotor adaptations in humans. They will open new scientific and clinical fields of study that will lead to the creation of motor rehabilitation paired with tVNS that can enhance rehabilitation outcomes in individuals with motor impairment. Demonstration of associated changes between central norepinephrine and neuromotor adaptations due to tVNS in non-disabled humans is a necessary step for applying tVNS to rehabilitation with the understanding of the underlying mechanism and for potentially using central norepinephrine as a predictor of tVNS efficacy in rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Men and women in the age range of 18-39 years will be recruited. All subjects will be healthy and right-handed. Subjects will match the ethnic distribution in the local community.

Exclusion Criteria:

* To ensure the safety associated with TMS and transcutaneous afferent vagus nerve stimulation, following adults will be excluded as in our previous studies (Buharin et al. 2013, 2014) and following the standard recommendations (Keel et al. 2001):

  1. Younger than 18 years old or older than 39 years old
  2. Left-handed
  3. Skilled use of hands (e.g. professional musician)
  4. High blood pressure (>140/90 mmHg)
  5. Had cardiovascular problems
  6. Obese (Body Mass Index: > 30 kg/m2)
  7. Had sensory deficits in your limb
  8. Had alcoholism
  9. Had psychiatric disorders
  10. Had an adverse reaction to TMS (a technique for non-invasive neural stimulation from the brain)
  11. Had a seizure (an abnormal phenomenon of the brain marked by temporary abnormal neuronal activity. Symptoms include involuntary changes in body movement or function, sensation, awareness, or behavior.)
  12. Someone in your family has epilepsy (recurrent seizures marking excessive synchronous neuronal activity in the brain)
  13. Had an EEG (measurement of the electrical activity of the brain through the use of surface electrodes placed on the scalp) for clinical diagnosis
  14. Had a stroke (the loss of brain function due to an interruption in the blood supply to the brain)
  15. Had a head injury (include neurosurgery) that required a visit to a hospital
  16. Suffer from frequent or severe headaches (e.g., migraine headaches within the last six months)
  17. Have any metal permanently in your head (outside the mouth) such as shrapnel, surgical clips, or fragments from welding or metal work. Piercings and other metals on your head are OK if they will be removed before the study.
  18. Have any implanted devices such as cardiac pacemakers (a medical device that uses electrical signals to regulate heart beat), medical pumps, or intra-cardiac lines
  19. Had any other brain-related condition
  20. Had any illness that caused brain injury (i.e. meningitis, aneurysm, brain tumor)
  21. Had severe disease such as cardiologic, pulmonary, renal, endocrinal (hyperthyroidism or hypothyroidism), gastrointestinal or others.
  22. Taking any medications other than over-the-counter medicine
  23. Suspect you might be pregnant (if woman)
  24. Have hearing problems, such as impaired hearing, tinnitus, etc.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2021-06-28 (Actual); Study Completion 2021-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Minoru Shinohara, PhD, Principal Investigator — Georgia Institute of Technology
Locations (1):
- Human Neuromuscular Physiology Lab, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from May 2019 to June 2021 through flyers posted in the classroom buildings and recreational buildings on the Georgia Tech campus.
Pre-assignment Details: There was no significant event in the study that occurred after participant enrollment.
Period: Overall Study
Arm/Group | Sham-tVNS to Ear Lobe | tVNS to Tragus
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham-tVNS to Ear Lobe | tVNS to Tragus | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 24
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 6 | 7 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 5 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 7 | 15
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Visuomotor Skill [Mean (Standard Deviation); unit: % of maximal voluntary contraction (MVC)] — The visuomotor skill was assessed with the root-mean-square error of the produced force against the target force, which was normalized to the maximal voluntary contraction force (MVC) of the finger and expressed in %MVC. A lower value is considered a smaller error and thus a better outcome.
  % of maximal voluntary contraction (MVC) | 1.89 (0.54) | 1.62 (0.56) | 1.76 (0.55)

OUTCOME MEASURES:

1. Primary Outcome: Visuomotor Skill
Description: Visuomotor skill was assessed with the amount of force error against the target trajectory. In the visuomotor task, subjects produced finger force against a force transducer to match a target trajectory as close as possible. The target was made of three low-frequency sinusoids with each sinusoid at different frequencies and amplitudes. This pattern spanned 20 s. The data in the middle 16 s were used for data analysis. For determining the visuomotor skill, the deviation of produced force from the target trajectory was calculated as the root-mean-square error. In this calculation, the difference between the target and produced force at each sampling point was squared, the squared values were summed across sampling points, and the squared root value of the summed value was determined and normalized to the maximal voluntary contraction (MVC) force. The data were expressed as the ratio of the baseline value (no unit). A lower value is considered a better outcome.
Time Frame: Day 1 (Baseline), Day 2 - 4, and Day 5 (Post)
Measure: Mean (Standard Deviation); unit: Ratio of the baseline value
Arm/Group | Sham-tVNS to Ear Lobe | tVNS to Tragus
Number analyzed (Participants) | 12 | 12
Ratio of the baseline value
  Day 1 (Baseline) | 1 (0) | 1 (0)
  Day 2 | 0.870 (0.213) | 0.969 (0.259)
  Day 3 | 0.616 (0.151) | 0.805 (0.198)
  Day 4 | 0.597 (0.215) | 0.683 (0.137)
  Day 5 (Post) | 0.551 (0.251) | 0.597 (0.149)
Statistical Analysis 1: Comparison: Sham-tVNS to Ear Lobe vs tVNS to Tragus; Test type: Superiority; p = 0.0096, ANOVA

2. Primary Outcome: Brain Excitability (MEP Amplitude)
Description: Brain excitability was assessed with motor evoked potential (MEP) amplitude of the resting first dorsal interosseus muscles as resting corticospinal excitability. Surface EMG electrodes were attached over the muscle in a belly-tendon configuration. Subjects received single-pulse TMS to evoke MEP in the muscle. MEP was obtained from the surface EMG using a high-gain EMG preamplifier. Peak-to-peak- amplitude of MEP in response to TMS were averaged across the intensities of 115-160% relative to the resting motor threshold. Additionally, maximal M-wave amplitude was obtained by stimulating the ulnar nerve that innervates the muscle. MEP amplitude was normalized to the maximal M-wave amplitude of the muscle, so it was expressed in % of maximal M-wave. A higher value is considered higher brain excitability and a better outcome.
Time Frame: Day 1 (Baseline) and Day 5 (Post)
Measure: Mean (Standard Deviation); unit: percentage of maximal M-wave
Arm/Group | Sham-tVNS to Ear Lobe | tVNS to Tragus
Number analyzed (Participants) | 12 | 12
percentage of maximal M-wave
  Day 1 (Baseline) before practice | 10.2 (6.4) | 13.2 (10.4)
  Day 1 (Baseline) after practice | 11.2 (6.8) | 17.7 (18.6)
  Day 5 (Post) before practice | 13.3 (19.9) | 11.0 (8.6)
  Day 5 (Post) after practice | 10.1 (6.9) | 11.8 (7.3)
Statistical Analysis 1: Comparison: Sham-tVNS to Ear Lobe vs tVNS to Tragus; Test type: Superiority; p = 0.764, ANOVA

3. Primary Outcome: Salivary Amylase Activity
Description: Central noradrenaline was assessed indirectly with salivary amylase activity. Saliva was sampled via salivette strips in the resting state before and after the training. Subjects were seated and rested for 5 minutes before sampling the samples. Collected saliva samples were immediately analyzed by using a dry-chemistry system automatically. Three saliva samples were analyzed and averaged across samples. Salivary amylase activity was measured and expressed in kU/I (kilo units per liter).
Time Frame: Day 3
Population: The number of participants is 11 (not 12) in each group because data were not obtained in one subject in the Sham-tVNS group and one subject in tVNS group due to technical difficulties during the measurement.
Measure: Mean (Standard Deviation); unit: kU/l
Arm/Group | Sham-tVNS to Ear Lobe | tVNS to Tragus
Number analyzed (Participants) | 11 | 11
kU/l
  Before intervention | 48.8 (25.1) | 46.0 (22.5)
  After intervention | 47.4 (15.7) | 52.4 (19.7)
Statistical Analysis 1: Comparison: Sham-tVNS to Ear Lobe vs tVNS to Tragus; Test type: Superiority; p = 0.446, ANOVA

ADVERSE EVENTS:
Time Frame: Up to one week
Arm/Group | Sham-tVNS to Ear Lobe | tVNS to Tragus
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-16): https://cdn.clinicaltrials.gov/large-docs/76/NCT03628976/Prot_SAP_001.pdf
  • Informed Consent Form (2021-04-16): https://cdn.clinicaltrials.gov/large-docs/76/NCT03628976/ICF_000.pdf